CLINICAL TRIAL: NCT06029075
Title: tACS Brain Neuromodulation for Sensory and Motor Recovery After Neurological Impairments
Brief Title: tACS for Neuropathic Pain Management After SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-22-0046 (Experiment 2)
Record Dates: First submitted 2023-05-10; First posted 2023-09-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Neuropathic Pain Management
Keywords: tACS; Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- "tACS Sham, tACS 10Hz, tACS 20Hz" experimental order (Experimental): 1. tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  2. tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  3. tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz
- "HD-tACS 20Hz, HD-tACS 10Hz, HD-tACS Sham" experimental order (Experimental): 1. tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  2. tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  3. tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz
- "HD-tACS 10Hz, HD-tACS 20Hz, HD-tACS Sham" experimental order (Experimental): 1. tACS 10Hz is a 10Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp or 20 or 40 minutes to entrain neuronal activity into 10Hz frequency patterns.
  2. tACS 20Hz is a 20Hz non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for 20 or 40 minutes to entrain neuronal activity into 20Hz frequency patterns.
  3. tACS Sham is a temporary non-invasive electrical stimulation that applies a weak oscillatory current to the brain through the scalp for up to 30 second, it is not designed to entrain neuronal activity into any external regulatory frequency patterns.
  Interventions: Device: tACS Sham; Device: tACS 10Hz; Device: tACS 20Hz

INTERVENTIONS:
Device: tACS Sham — Sham tACS will applied to the brain through the scalp for 20 minutes.
Device: tACS 10Hz — 10Hz tACS will applied to the brain through the scalp for 20 minutes.
Device: tACS 20Hz — 20Hz tACS will applied to the brain through the scalp for 20 minutes.

SUMMARY:
The overall goal is to investigate the effectiveness of a novel intervention - transcranial alternating current stimulation (tACS) for neuropathic pain management in people after spinal cord injury.

ELIGIBILITY:
Inclusion/exclusion criteria for SCI subjects

Inclusion criteria: A patient who

1. has neuropathic pain after traumatic spinal cord injury or amputation or brain injury;
2. has chronic pain, >3 months;
3. is between 18 to 75 years of age;
4. is stable on oral pain medications at least two weeks. Patients are allowed to continue their pain medications, i.e., no change in pain medications.

NOTE: we plan to begin the study with the spinal cord injury (SCI) subject population as a cohort first, then expand to other subject populations

Exclusion criteria: Patients will be excluded if they

1. are currently adjusting oral pain medications for their neuropathic pain;
2. have pain, but not neuropathic, e.g., from inflammation at the incision wound of the residual limb or neuroma;
3. have a pacemaker metal implants or supplemental oxygen;
4. have amputation in their arm(s);
5. fail to have a motor contraction in the arm muscles with TMS;
6. are not able to follow commands, or to give consent;
7. have asthma or other pulmonary disease;
8. are not medically stable;
9. have preexisting psychiatric disorders;
10. alcohol or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain scale (visual analogue scale, VAS) measurement | Change of VAS 5 minutes before and after the tACS intervention will be measured.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Heart rate variability (HRV) measurement | Change of HRV 10-15 minutes before and after the tACS intervention will be measured.
  Heart rate variability (HRV) is the fluctuation in the time intervals between adjacent heartbeats (1). HRV indexes neurocardiac function and is generated by heart-brain interactions and dynamic non-linear autonomic nervous system (ANS) processes. HRV will be used as a surrogate assessment for autonomic nerve system

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, Ph.D, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No